CLINICAL TRIAL: NCT00906919
Title: The Effectiveness of Diabetes Patient Education and Self-Management Education in Persons With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Vancouver Foundation (Other)
Responsible Party: Patrick McGowan, PhD, University of Victoria - Centre on Aging
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BCM03-0095
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: self-efficacy; health behavior; patient education; health education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Behavior; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular diabetes patient education (Active Comparator): Regular professionally-led diabetes patient education
  Interventions: Behavioral: Regular diabetes patient education
- Augmented Diabetes Patient Education (Experimental): Regular professionally-led diabetes patient education augmented by participation in the Stanford Chronic Disease Self-Management Program
  Interventions: Behavioral: Augmented diabetes patient education

INTERVENTIONS:
Behavioral: Regular diabetes patient education — Professionally-led diabetes patient education delivered by health professionals over a two day period
  Arms: Regular diabetes patient education
Behavioral: Augmented diabetes patient education — Professionally-led diabetes patient education led by nurse and dietitian over a two day period augmented by participation in the Stanford Chronic Disease Self-Management Program. This program takes place for 2 1/2 hours per week for six consecutive weeks.
  Arms: Augmented Diabetes Patient Education

SUMMARY:
The goal of this randomized controlled trial is to determine if greater effectiveness can be achieved by the addition of lay-led self-management patient education to regular professionally-led diabetes patient education in comparison to regular professionally-led diabetes patient education only.

DETAILED DESCRIPTION:
In the current health care environment, it is unacceptable for patient education programs to merely provide information. Rather, educational programs must concentrate on behavior change and on supporting patients to become more confident and motivated in participating in managing their health. Persons with type 2 diabetes attending a Diabetes Education Centre will be assigned to either a group that receives regular professionally-led diabetes patient education (control group) or to to a group that receives regular professionally-led diabetes patient education augmented by lay-led self-management education i.e., the Stanford six-session Chronic Disease Self-Management Program (experimental group). Data will be collected at two points in time (0 and 6 months). Outcome measures will show if participants who receive self-management training in addition to regular patient education are able to:manage their diabetes more effectively; engage in the specific behaviors that keep the condition from worsening; achieve more control over their condition; and use the health care system more effectively.

ELIGIBILITY:
Inclusion Criteria:

* adults with type 2 diabetes

Exclusion Criteria:

* cognitive impairment
* unable to speak English

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2004-04; Primary Completion 2007-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
A1C | 6 months

SECONDARY OUTCOMES:
Self-management behaviors | 6 months
Self-efficacy levels | 6 months
Health status | 6 months
Cholesterol levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T McGowan, PhD, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria - Centre on Aging (Ladner Office), Suite 210, 4907 Chisholm Street, Delta, British Columbia, Canada